CLINICAL TRIAL: NCT02107222
Title: A Multicenter Randomized Control Trial (RCT) to Determine Safety and Efficacy of PALP™ for ECCO2-R in Conjunction With Liberation From Mechanical Ventilation (MV) Compared to MV Alone in COPD Exacerbation and Respiratory Failure
Brief Title: The PALP™-COPD Trial (Low-Flow CO2-Removal (ECCO2-R) in Exacerbated COPD)
Acronym: PALP-COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This action is an internal decision that was not made because of any pending regulatory action for these products.
Sponsor: Maquet Cardiopulmonary GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAQ/COPD/PALP/2012
Record Dates: First submitted 2014-03-28; First posted 2014-04-08 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: COPD; Exacerbation; invasive ventilation; CO2-Removal
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mechanical ventilation (MV) (No Intervention): mechanical ventilation according to guidelines
- MV + ECCO2-R(PALP-Device/MaquetCP) (Experimental): MV according to the guidelines plus CO2-Removal with PALP
  Interventions: Device: CO2-Removal (PALP-Device/MaquetCP)

INTERVENTIONS:
Device: CO2-Removal (PALP-Device/MaquetCP) — extracorporeal circuit to remove CO2 out of the blood
  Arms: MV + ECCO2-R(PALP-Device/MaquetCP)

SUMMARY:
A Multicenter, Randomized, Controlled Trial to Determine Safety and Efficacy of Pump Assisted Lung Protection (PALP™) for Low Flow Carbon Dioxide (CO2) Removal in Conjunction with Liberation from Mechanical Ventilation Compared to Mechanical Ventilation Alone in Patients with COPD Exacerbation and Respiratory Failure

DETAILED DESCRIPTION:
Primary Study Objectives

• To evaluate the clinical effect of PALP™ in reducing the time on invasive ventilation in patients with an exacerbation of COPD requiring invasive mechanical ventilation.

Secondary Study Objectives

* To evaluate the safety and tolerability of PALP™ in patients with an exacerbation of COPD requiring invasive mechanical ventilation.
* To determine if rates of adverse events (AEs) are reduced in patients who receive PALP™ and invasive mechanical ventilation vs invasive mechanical ventilation alone.
* To determine mortality rates in patients who receive PALP™ and invasive mechanical ventilation vs invasive mechanical ventilation alone.
* To determine if PALP™ will effectively reduce the number of subsequent acute decompensations requiring hospital admission for ventilatory support (invasive or noninvasive).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, and ≥40 years of age
2. Known history of COPD
3. Currently experiencing an exacerbation of COPD
4. P/F ratio >150 mmHg
5. Currently endotracheally intubated and requiring invasive mechanical ventilation (must have been on invasive mechanical ventilation for 24-48 hours)
6. Able to tolerate large bore intravenous (IV) cannulation required for proper operation of study device
7. For female patients of child-bearing potential, a negative urine or serum pregnancy test at screening; all female patients will be considered of child-bearing potential unless they are post menopausal for at least 1 year or have been surgically sterilized (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)
8. Written informed consent obtained according to local regulations; or, if unable to provide written informed consent due to incapacitation, a legally authorized representative is able to provide written informed consent on behalf of the patient

Exclusion Criteria:

1. Any end-stage medical conditions with expected survival <6 months
2. Tracheostomy
3. Unable to provide central venous access
4. Acute brain injury
5. Any legally authorized document(s) that may restrict aggressive medical management such as "Do Not Resuscitate," "Do Not Intubate," etc.
6. Risk of bleeding or clotting such as:

   * Known bleeding diathesis or abnormal clotting
   * Recent or current use of medications known to increase risk of bleeding
7. Screening platelet count of <75,000/mm3 or international normalized ratio (INR) >1.5 or activated partial thromboplastin time (aPTT) >1.5 times the upper limit of normal (ULN) range for their respective laboratory values
8. Any recognized contra indications to systemic anticoagulation therapy or use of heparin
9. Body mass index (BMI) >35
10. Any form of chronic hyperventilation not related to COPD
11. Hemodynamic instability or requiring significant vasopressor support
12. Cardiogenic or noncardiogenic pulmonary edema as the primary reason for respiratory failure
13. High risk cardiac conditions
14. Oxygen tension in arterial blood (PaO2) <50 mmHg via arterial blood gas (ABG) or any condition in which hypoxemia is a significant component of the respiratory failure
15. Any other medical cause for acute respiratory failure not directly related to a COPD exacerbation
16. Use of or treatment with an investigational drug, therapy, or device within 1 month (30 days) of baseline
17. Female patients who are pregnant or breastfeeding
18. Patients who are immuno-compromised
19. Current active malignancy or history of malignancy within the past 5 years
20. Patients in chronic dialysis
21. Patients requiring extra-corporeal life support (ECLS) as a bridge to transplant
22. Patients who, in the opinion of the investigator, would not be able to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Difference in time of mechanical ventilation | 720 hours
  • To evaluate the clinical effect of PALP™ in reducing the time on invasive ventilation in patients with an exacerbation of COPD requiring invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Marco V Ranieri, MD PhD, Principal Investigator — Investigational institution
Locations (1):
- MAQUET Cardiopulmonary AG, Rastatt, Germany

REFERENCES:
- [Result] Abrams DC, Brenner K, Burkart KM, Agerstrand CL, Thomashow BM, Bacchetta M, Brodie D. Pilot study of extracorporeal carbon dioxide removal to facilitate extubation and ambulation in exacerbations of chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2013 Aug;10(4):307-14. doi: 10.1513/AnnalsATS.201301-021OC. PMID 23952848